CLINICAL TRIAL: NCT05207332
Title: The Effect of a Vegan Alginate Product on Athletes Recovery and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Bendix Jeppesen (Other)
Collaborators: Future Food Innovation (Industry)
Responsible Party: Sponsor-Investigator, Per Bendix Jeppesen, Associate professor, Ph.D., Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: VEGSPORT
Record Dates: First submitted 2019-03-14; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Athletic Performance
MeSH Terms: interventions — CVS 1123

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan product (Experimental)
  Interventions: Dietary Supplement: CHO+PRO
- Control (Active Comparator)
  Interventions: Dietary Supplement: CHO

INTERVENTIONS:
Dietary Supplement: CHO+PRO — A vegan product containing carbohydrate and protein
  Arms: Vegan product
Dietary Supplement: CHO — containing carbohydrate
  Arms: Control

SUMMARY:
The feeding strategies during recovery are essential to optimize a subsequent performance. Carbohydrate is a major fuel source during exercise as it has been shown to maintain high rates of carbohydrate oxidation. Protein intake in combination with carbohydrate have been shown to increase Amino acid bioavailability and may alter physiologic responses during exercise, which may be relevant to endurance performance. The goal of this study is to assess the effect of a new developed vegan product on athletes recovery and subsequent performance.

ELIGIBILITY:
Inclusion Criteria:

* males between 18-50 years of age
* moderate to trained individuals with a VO2max > 50 ml/min/kg

Exclusion Criteria:

* persons diagnosed with metabolic diseases (i.e. Type 2 Diabetes) which relates to the carbohydrate metabolism.
* persons ingesting prescribed drugs/medicin, supplements or a special diet (i.e. low carbohydrate), which might affect the glykogen synthesis and/or performance.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Performance | Aprox. 120 minutes
  Time-to-exhaustion. Measured by the duration of high intensity exercise performed to exhaustion.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Denmark